CLINICAL TRIAL: NCT05933928
Title: The Effect of Simulation-Based Electronic Fetal Monitoring Training on Self-Efficacy-Efficacy and Anxiety Levels of Midwifery Students
Brief Title: The Effect of Simulation-based Electronic Fetal Monitoring Training on Midwifery Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBÜ-AYDINKARTAL-004
Record Dates: First submitted 2023-06-24; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Fetal Monitoring
Keywords: EFM; midwifery students; simulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind quasi-experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (High validity simulation application group) (n:40) (Experimental): Practices will be carried out with the students in the intervention group with the "NOELLA Birth Simulator", which is a high-reality simulator located in the Simulation laboratory of the Department of Midwifery of the Faculty of Health Sciences of Hamidiye. A simulator will be practiced with a separate scenario including early, late, variable deceleration, reactive, sinusoidal and non-reactive trace interpretation and intervention.
  Interventions: Other: Simulation-based electronic fetal monitoring training
- Control group (Case-based teaching technique group) (n:40) (No Intervention): To the control group students; Cases on early, late, variable deceleration, reactive, sinusoidal and non-reactive tracing will be prepared by dividing into groups of 5 people. Semi-structured cases will be evaluated and clinical intervention will be discussed with group work. Practice will be done in the basic skills laboratory of the midwifery department.

INTERVENTIONS:
Other: Simulation-based electronic fetal monitoring training — Practices will be carried out with the students in the intervention group with the "NOELLA Birth Simulator", which is a high-reality simulator located in the Simulation laboratory of the Department of Midwifery of the Faculty of Health Sciences of Hamidiye. A simulator will be practiced with a separate scenario including early, late, variable deceleration, reactive, sinusoidal and non-reactive trace interpretation and intervention.
  Arms: İntervention group (High validity simulation application group) (n:40)

SUMMARY:
This study was planned to determine the effect of scenario-based high-fidelity electronic fetal monitoring simulation method on midwifery students' self-efficacy-efficacy and situational anxiety levels. The study was planned as a randomized controlled experimental study. This RCT will be administered following the CONSORT 2010 guidelines. Midwifery students will be given information about the introduction of the simulator and the model, the flow chart of the training plan, the content of the training plan, the environment, the locations of the materials. 40 students selected for the intervention group will be given high-fidelity simulator and information on case-based learning will be given to 40 students selected for the training and control group. "State Anxiety Inventory" and "Self-Efficacy-Efficacy Scale" will be applied as a pre-test after the briefing. High-fidelity simulator application training will be applied to the intervention group students, accompanied by a scenario, and case-based learning method will be applied to the control group students. After the training, "State Anxiety Inventory", "Self-Efficacy-Efficacy Scale" and "Satisfaction with Educational Methods Questionnaire" will be administered to all students. Three months after the training, the "State Anxiety Inventory" and "Self-Efficacy-Efficacy Scale" will be administered to the students again.

DETAILED DESCRIPTION:
It was planned to determine the effect of scenario-based high-reality Electronic Fetal Monitoring (EFM) simulation method on midwifery students' self-efficacy, competence and situational anxiety levels.

The population of the research will be Health Sciences University Hamidiye Health Sciences Faculty Midwifery Department 3rd year students (N:80). In this study, which was planned as a quasi-experimental pre- and post-test design and with a control group, all students who are actively studying in the 3rd year of the midwifery department, whose sample selection was not made, will form the scope of the research, and individuals who volunteered to participate in the study will form the sample of the research.

The students who volunteered to participate in the study will be assigned to the intervention and control groups with a computer-assisted simple random sampling method. Computer-assisted randomization will be used in the study, and random assignment will be made to the intervention and control groups by entering the number of cases through the program whose URL is https://www.randomizer.org. After 4 hours of theoretical training on EFM application and interpretation are given to all students, intervention group students will be given a scenario-accompanied high-validity simulation laboratory application, and control group students will be given only case-based learning technique.

All groups will be informed before the applications. In this context, a question-and-answer session will be held by giving information about the applications to be made regarding the research. Students will be given information about the introduction of the simulator and the model, the flow chart of the training plan, the content of the training plan, the environment, the locations of the materials. 40 students selected for the intervention group will be given high-fidelity simulator and information on case-based learning will be given to 40 students selected for the training and control group. Before the application, all groups will be given theoretical information about electronic fetal monitoring for 4 hours with a power point presentation. "State Anxiety Inventory" and "Self-Efficacy Scale" will be applied as a pre-test after the briefing. High-fidelity simulator application training will be applied to the intervention group students, accompanied by a scenario, and case-based learning method will be applied to the control group students. After the training, "State Anxiety Inventory", "Self-Efficacy Scale" and "Satisfaction with Educational Methods Questionnaire" will be administered to all students. Three months after the training, the "State Anxiety Inventory" and "Self-Efficacy Scale" will be administered to the students again.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research.
* Being a third year student at SBU, Hamidiye Faculty of Health Sciences, Midwifery Department.

Exclusion Criteria:

* Not volunteering to participate in the research.
* Not to be a third year student at the Faculty of Health Sciences, Hamidiye, Department of Midwifery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | One hour before the education
  In this form, which was created by the researchers based on the literature, participants' age, high school they graduated from, willingly choosing the profession, feeling of belonging to the profession, etc. questions are included.
State-Trait Anxiety Inventory | One hour before the education
  The scale consists of two subscales, continuous and state, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how the individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how the individual feels independently of the situation and conditions. The scores obtained from the scale theoretically vary between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
Self-Efficacy Scale | One hour before the education
  The scale, which does not belong to any subjective domain, measures the perception of general self-efficacy and efficacy. The Self-Efficacy Scale is structured as a 5-point Likert-type scale consisting of 23 items, and a minimum of 23 and a maximum of 115 points can be obtained from the scale. For each item on the scale, one of the options 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well, is based on the score given for each item. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 on the scale are scored in the opposite direction. An increase in the total score that can be obtained from the scale indicates that the general self-efficacy perception is high.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | After education
  The scale consists of two subscales, continuous and state, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how the individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how the individual feels independently of the situation and conditions. The scores obtained from the scale theoretically vary between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
Self-Efficacy Scale | After education
  The scale, which does not belong to any subjective domain, measures the perception of general self-efficacy and efficacy. The Self-Efficacy Scale is structured as a 5-point Likert-type scale consisting of 23 items, and a minimum of 23 and a maximum of 115 points can be obtained from the scale. For each item on the scale, one of the options 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well, is based on the score given for each item. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 on the scale are scored in the opposite direction. An increase in the total score that can be obtained from the scale indicates that the general self-efficacy perception is high.
Satisfaction Survey with Training Methods | After education
  The questionnaire consists of 16 propositions. One of these propositions is the proposition "I am satisfied with this education method in general", which questions the state of being satisfied with the education. Other propositions were formed from propositions aiming to determine the views of the education method in general about the contribution of the education method to the learning and professional life of the student. Each proposition is scored on a 5-point Likert scale (1-strongly disagree, 5-strongly agree). It is determined that as the scale score average increases, students' satisfaction with the education method increases, and as the scale score average decreases, their satisfaction with the education method decreases.

OTHER OUTCOMES:
State-Trait Anxiety Inventory | Three months after the education
  The scale consists of two subscales, continuous and state, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how the individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how the individual feels independently of the situation and conditions. The scores obtained from the scale theoretically vary between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
Self-Efficacy Scale | Three months after the education
  The scale, which does not belong to any subjective domain, measures the perception of general self-efficacy and efficacy. The Self-Efficacy Scale is structured as a 5-point Likert-type scale consisting of 23 items, and a minimum of 23 and a maximum of 115 points can be obtained from the scale. For each item on the scale, one of the options 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well, is based on the score given for each item. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 on the scale are scored in the opposite direction. An increase in the total score that can be obtained from the scale indicates that the general self-efficacy perception is high.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Aydın Kartal Assoc. Prof. Dr., Principal Investigator — Saglik Bilimleri Universitesi; Aleyna Bulut Research Assistant, Study Chair — Saglik Bilimleri Universitesi; Sema Aker Research Assistant, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No